CLINICAL TRIAL: NCT03073798
Title: The Effectiveness of Roflumilast in Improving Mucociliary Clearance in Patients With COPD and Chronic Bronchitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00078710
Record Dates: First submitted 2017-03-02; First posted 2017-03-08 (Actual); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: COPD; Chronic Bronchitis; Emphysema
Keywords: Lung Disease; Breathing Difficulty; Smoking; Mucociliary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Lung Diseases; Dyspnea; Smoking | interventions — Roflumilast; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medication (Active Comparator): Roflumilast. 500 mcg of Roflumilast daily for 4 weeks, then there will be a 4 week wash-out phase (no medication) and a second 4 week period of placebo.
  Interventions: Drug: Roflumilast; Drug: Placebo
- Placebo (Placebo Comparator): Placebo. 500 mcg of Placebo daily for 4 weeks, then there will be a 4 week wash-out phase (no medication) and a second 4 week period of Roflumilast
  Interventions: Drug: Roflumilast; Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 mcg of Roflumilast which is a prescription medicine used in adults with severe COPD to decrease the number of flare-ups or the worsening of COPD symptoms
  Other Names: Daliresp
Drug: Placebo — 500 mcg of placebo is used
  Other Names: Sugar Pill

SUMMARY:
Specific Aim: To determine the effectiveness of Roflumilast in improving i) whole right lung and ii) peripheral right lung mucociliary clearance (MCC) in patients with COPD and chronic bronchitis.

Hypothesis: Roflumilast increases mucociliary clearance in patients with chronic bronchitis.

Study Design: This will be a double-blinded, cross-over randomized controlled trial with 1:1 randomization of 20 individuals with chronic bronchitis. Subjects will undergo baseline MCC then will be randomized to either roflumilast or placebo x 4 weeks, then there will be a 4 week wash-out phase and a second 4 week period of roflumilast/placebo depending on initial randomization. MCC will be conducted at baseline and at the end of each 4 week medication phase.

DETAILED DESCRIPTION:
The purpose of this study is to investigate how well Roflumilast improves mucociliary clearance in people with chronic bronchitis. Several studies show that roflumilast may modulate (change) mucociliary function. This study is designed to determine if these favorable effects lead to improved mucociliary clearance (MCC) in people with chronic bronchitis, thereby, reducing the potential for acute infections and hospitalizations. Daliresp® (roflumilast) is a drug currently marketed (approved by the U.S. Food and Drug Administration (FDA) for use in humans) in the U.S. and is indicated (used) for treatment of people with severe COPD to treat the symptoms of cough and excess mucous linked to chronic bronchitis. Roflumilast is used to reduce the risk (chance) of COPD exacerbations (increase in symptoms such as cough, mucus secretions, and shortness of breath, that can be life threatening and reduces the ability to breathe) linked to chronic bronchitis (swelling of the airways in the lungs). Roflumilast is FDA approved to decrease the number of flare-ups of chronic obstructive pulmonary disease (COPD) in patients with severe COPD with chronic bronchitis and a history of flare-ups. The exact way Roflumilast does this is not known. Although Roflumilast is an FDA approved drug, in this study the drug is not being used for its FDA-approved indication.

If you agree to be in this study, you will receive no new COPD treatment other than the drugs provided for the study. You will also be given a tablet to take once a day, which will be placebo for at least part of the study. A placebo is a substance that looks like the study drug but that contains no active ingredients.

The study is a double-blind study. Double-blind means that neither you nor the study doctor will know which study regimen (roflumilast or placebo) you are receiving throughout the study. However, this information can be made available if medically necessary and as determined by the participant's study. You will undergo baseline mucociliary Clearance (MCC) Measurements then will be randomized (by chance, like the flip of a coin) to receive either roflumilast or placebo for 4 weeks, then there will be a 4 week wash-out phase, and a second 4 week period of roflumilast/placebo depending on initial randomization. Mucociliary Clearance (MCC) Measurements will be conducted at the beginning and at the end of each 4 week study regimen phase. You will be in the study for about 12 weeks and there will be up to 12 visits. At baseline, and prior to each MCC Procedure, you will have health assessments which may include Physical Examination, Health and Demographic Interview, Exhaled Carbon Monoxide (eCO) Testing, Spirometry (Breathing Test), Expectorated Sputum Collection, Pregnancy Testing and Mucociliary Clearance (MCC) Measurements.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of COPD
* Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) ≤70%
* FEV1 (% predicted) ≥40 % AND ≤ 70%,
* Tobacco exposure ≥ 10 pack-years,
* Chronic cough and sputum production
* At least one COPD exacerbation requiring systemic glucocorticosteroids or treatment in hospital, or both, in the previous year
* Not suffering from any concomitant disease that might interfere with study procedures or evaluations.

Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticosteroids and/or antibiotics not stopped at least 4 weeks prior to the baseline visit V0
* Lower respiratory tract infection not resolved 4 weeks prior to the baseline visit V0
* Diagnosis of asthma and/or other relevant lung disease (e.g. history of bronchiectasis, cystic fibrosis, bronchiolitis, lung resection, lung cancer, interstitial lung disease [e.g. fibrosis, silicosis, sarcoidosis], and active tuberculosis
* Known alpha-1-antitrypsin deficiency
* Known infection with HIV and/or active hepatitis
* Pregnancy or women of childbearing potential not using or willing to continue using a medically reliable method of contraception for the entire study period
* Suspected hypersensitivity to the study medication (roflumilast).
* Use of mucolytics within the last 4 weeks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hansel, MD MPH, Principal Investigator — Jonhs Hopkins University; Beth Laube, PhD, Principal Investigator — Jonhs Hopkins University

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Subjects underwent baseline MCC, then first received Roflumilast 500 mcg daily for 4 weeks. After a washout period of 4 weeks, they then received Placebo 500 mcg for an additional 4 weeks.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Roflumilast. 500 mcg of Roflumilast daily for 4 weeks, then there will be a 4 week wash-out phase (no medication) and a second 4 week period of placebo.
  Roflumilast: 500 mcg of Roflumilast which is a prescription medicine used in adults with severe Chronic Obstructive Pulmonary Disease (COPD) to decrease the number of flare-ups or the worsening of COPD symptoms
  Placebo: 500 mcg of placebo is used
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mucociliary Clearance (MCC) Between Visit 1A and Visit 2A
Description: Measurements of MCC (Mucociliary clearance) will be obtained using a large-field-of-view 2D gamma camera (Siemens Orbiter) following inhalation of a radioaerosol containing a gamma emitting isotope 99mtechnetium (99mTc)-sulfur-colloid. The total exposure to radiation from procedures associated with the MCC studies is similar to that of a chest x-ray and is much less than the 0.3 rem that the average person in the United States gets each year from natural sources like the sun, outer space, air, food, and soil.
  After inhaling (0 time point) an aerosol generated from a saline solution containing the radioisotope 99mtechnetium (99mTc)-sulfur-colloid (radioaerosol), subjects will sit with their back to a gamma camera. The gamma camera will acquire an image of where the isotopic marker initially deposits in the right lung at time 0 and how much remains in the lungs at the specified time point and will be measured in change of %/min from 0 min time point.
Time Frame: Change from 0 to 30 minutes
Population: Data was not collected for all participants in this outcome measure due to lack of follow-up, patient withdrawal from the study, and an adverse event.
Measure: Mean (Standard Deviation); unit: percentage difference of MCC
Groups:
- All Roflumilast MCC: Taking into account the washout period and crossover design of this study, we are presenting the results to reflect all of the MCC studies done while the participants were on roflumilast.
- All Placebo MCC: Taking into account the washout period and crossover design of this study, we are presenting the results to reflect all of the MCC studies done while the participants were on placebo.
Arm/Group | All Roflumilast MCC | All Placebo MCC
Number analyzed (Participants) | 9 | 10
percentage difference of MCC | -1.50 (3.76) | -0.70 (4.71)

2. Primary Outcome: Difference in Mucociliary Clearance (MCC) Between Visit 1A and Visit 2A
Description: as for outcome 1
Time Frame: Change from 0 to 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage difference of MCC
Arm/Group | All Roflumilast MCC | All Placebo MCC
Number analyzed (Participants) | 9 | 10
percentage difference of MCC | -2.18 (5.17) | 0.13 (5.81)

3. Primary Outcome: Difference in Mucociliary Clearance (MCC) Between Visit 1A and Visit 2A
Description: as for outcome 1
Time Frame: Change from 0 to 90 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage difference of MCC
Arm/Group | All Roflumilast MCC | All Placebo MCC
Number analyzed (Participants) | 9 | 10
percentage difference of MCC | -1.31 (7.77) | 0.52 (6.63)

4. Primary Outcome: Difference in Mucociliary Clearance (MCC) Between Visit 1B and Visit 2B
Description: as for outcome 1
Time Frame: Change from 0 min to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage difference of MCC
Arm/Group | All Roflumilast MCC | All Placebo MCC
Number analyzed (Participants) | 9 | 10
percentage difference of MCC | -0.13 (12.87) | 6.93 (18.50)

ADVERSE EVENTS:
Groups:
- All Participants: Subjects underwent baseline MCC, then first received Roflumilast 500 mcg daily for 4 weeks. After a washout period of 4 weeks, they then received Placebo 500 mcg for an additional 4 weeks.
  MCC was conducted at baseline and at the end of each 4 week medication phase.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=12)
Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One participant had a pulmonary exacerbation prior to drug administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes